CLINICAL TRIAL: NCT06946030
Title: The Relationship Between Ocular Pseudoexfoliation Syndrome and Carpal Tunnel Syndrome
Brief Title: Pseudoexfoliation and Carpal Tunnel Study
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Physical Medicine & Rehabilitation Specialist, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-05
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-04

CONDITIONS: Pseudoexfoliation Syndrome; Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome (CTS); pseudoexfoliation syndrome; Biochemical marker
MeSH Terms: conditions — Exfoliation Syndrome; Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pseudoexfoliation Group: Patients will be selected from among those diagnosed with Pseudoexfoliation Syndrome (PES). Patients who are diagnosed with PES during routine eye examination will be informed about the study, and if they agree to participate, detailed informed consent will be obtained. EMG will be performed on the same day for consenting patients to evaluate whether they have Carpal Tunnel Syndrome (CTS).
- Control Group: Control group will be selected from among patients who present to physical therapy outpatient clinics with complaints such as mechanical back, knee, or hip pain, without any symptoms or findings suggestive of CTS, and matched for age and sex ratio. Patients who will constitute the control group will also be informed about the study, and detailed informed consent will be obtained from those who agree to participate. Subsequently, EMG examination will be performed on the same day to evaluate the presence of CTS.

SUMMARY:
Investigation of the Association Between Ocular Pseudoexfoliation Syndrome (PES) and Carpal Tunnel Syndrome (CTS) with Biochemical Markers. To study the frequency of concurrent CTS and PES, and to analyze the association between PES and CTS severity.

DETAILED DESCRIPTION:
Pseudoexfoliation syndrome (PES), first described by Lindberg in 1917, is a relatively common systemic disorder. While it primarily affects ocular tissue through gradual accumulation of fibrogranular material in the anterior segment of the eye, it can be observed in any other tissue. The chemical composition of the accumulated material is still not fully understood. Abnormal metabolism and overproduction of glycosaminoglycans are thought to play a key role. PES is commonly seen in males and individuals over 60 years of age, with incidence varying according to race and geographical characteristics.

This syndrome manifests itself with flaking at the pupillary margin and anterior lens capsule, increased pigmentation in the trabecular meshwork, and open-angle glaucoma. In PES, extracellular matrix deposits, exfoliative material, and amyloid accumulations have been demonstrated in other organs as well. Relationships between PES and systemic diseases such as diabetes mellitus, ischemic heart diseases, cerebrovascular diseases, and hypertension have been reported.

PES, defined as a neurodegenerative disease, has also been reported to be associated with Alzheimer's disease. It has been reported that PES affects peripheral nerves and has a direct relationship with carpal tunnel syndrome (CTS).

CTS is a condition resulting from compression of the median nerve in the carpal tunnel at the wrist and is the most common entrapment neuropathy. CTS is most commonly seen in the 3rd-5th decades and is three times more common in women than men. Most cases are idiopathic where the cause cannot be determined. While repetitive trauma is most commonly blamed in the etiology, some systemic diseases, primarily obesity, diabetes mellitus (DM), and rheumatoid arthritis (RA), are reported to play a role.

High body mass index (BMI) is an important risk factor in the development of CTS. A positive correlation between BMI and CTS severity has been reported. It has been found that CTS is more common and more severe in patients with metabolic syndrome, an endocrinopathy characterized by abdominal obesity, atherogenic dyslipidemia, high blood pressure, insulin resistance or glucose intolerance, and prothrombotic and proinflammatory states. Dyslipidemia encountered in metabolic syndrome is characterized by high triglycerides and low HDL. Dyslipidemia is reported to make a significant contribution to peripheral nerve deterioration.

Dyslipidemia has also been reported in PES patients. Although a specific pathogenesis in PES is still unknown, hypoxia, ischemia, chronic inflammation, oxidative stress, and decreased cellular defense are emphasized. In PES, increased homocysteine levels along with decreased levels of vitamin B12 and folate, which are cofactors in homocysteine metabolism, have been reported. Study results regarding the relationship between vitamin B12 and CTS are contradictory.

Our aim in this study is to investigate the frequency of co-occurrence of PES and CTS. Literature information about the association of PES and CTS is limited. The purpose of this study is to make a new evaluation on this subject and contribute to the literature. Thus, we believe we can reach data that will lay the groundwork for more comprehensive future research focused on common pathophysiology for these two syndromes whose etiopathogenesis has not been fully elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-90
* Having been diagnosed with PES during routine eye examination

Exclusion Criteria:

* History of major hand-wrist trauma or surgical intervention
* Acromegaly
* Presence of any structural abnormality in bone structure
* Pregnancy
* Diabetes mellitus
* Gout
* Rheumatoid arthritis
* Connective tissue disease
* Acromegaly
* Thoracic outlet syndrome
* Brachial plexopathy
* Cervical disc herniation
* Presence of cardiac pacemaker
* Steroid users
* Thyroid disease
* Repetitive hand operations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case group participants will be selected from patients diagnosed with PES during eye examination. After informed consent, EMG will be performed to evaluate for CTS. Boston CTS Questionnaire will assess symptom severity in CTS-positive patients. Demographics, comorbidities, EMG and questionnaire results will be recorded. Control group will consist of age/gender-matched patients with mechanical back, knee, or hip pain without CTS symptoms. They will also undergo EMG after consent. All demographic data, comorbidities, and EMG results will be documented for both groups.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Electromyography (EMG) | up to 12 weeks
  Electromyography (EMG) is an examination method that measures the electrical conduction function of nerves using linear electrical current at an intensity that will not cause excessive discomfort to the patient. For this purpose, low-intensity electrical current is applied to the fingers and skin areas over the nerves, and this current is collected and measured by computerized devices from another part of the nerve or skin. Thus, it is determined whether the nerve is functioning properly.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ) | up to 12 weeks
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ); Boston Questionnaire Form (BQF), consists of a total of 19 questions. It includes 11 questions to assess symptom severity and 8 questions to evaluate functional capacity. Responses are multiple-choice and are scored from a minimum of one to a maximum of five points for each question. One point corresponds to the mildest symptom or best functional status, while five points correspond to the most severe symptom or worst functional status. A high average score indicates severe complaints or inadequate functional capacity. The symptom severity score is the total score obtained from 11 questions. The average symptom severity score is calculated by dividing the total score obtained from 11 questions by eleven. The functional capacity score is the total score obtained from eight questions. The average functional capacity score (AFCS) is obtained by dividing this score by eight.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The collected individual patient data contains sensitive personal health information protected by privacy regulations. Due to ethical considerations and patient confidentiality requirements specified in our informed consent protocol, we are unable to share the raw individual patient data with other researchers. However, aggregated and anonymized statistical results will be made available through scientific publication.

REFERENCES:
- [Background] Tarim B. The role of serum biomarkers in determining systemic inflammation and cardiovascular risk in pseudoexfoliation syndrome. Int Ophthalmol. 2024 Dec 19;45(1):15. doi: 10.1007/s10792-024-03382-5. PMID 39699776
- [Background] Otelea MR, Nartea R, Popescu FG, Covaleov A, Mitoiu BI, Nica AS. The Pathological Links between Adiposity and the Carpal Tunnel Syndrome. Curr Issues Mol Biol. 2022 Jun 8;44(6):2646-2663. doi: 10.3390/cimb44060181. PMID 35735622
- [Background] Malakootian M, Soveizi M, Gholipour A, Oveisee M. Pathophysiology, Diagnosis, Treatment, and Genetics of Carpal Tunnel Syndrome: A Review. Cell Mol Neurobiol. 2023 Jul;43(5):1817-1831. doi: 10.1007/s10571-022-01297-2. Epub 2022 Oct 10. PMID 36217059
- [Background] Shahriari M, Karimzadeh A, Esmaily H, Rezanejad S, Nikkhah H, Yadgari M, Pourhoseingholi A. Electrodiagnostic signs of carpal tunnel syndrome in ocular pseudoexfoliation syndrome. Int Ophthalmol. 2022 Sep;42(9):2749-2755. doi: 10.1007/s10792-022-02264-y. Epub 2022 Apr 27. PMID 35478398
- [Background] Padhy B, Alone DP. Is pseudoexfoliation glaucoma a neurodegenerative disorder? J Biosci. 2021;46:97. PMID 34785624
- [Background] Patil VR, Vallabha K, Wali K. Systemic Vascular Parameters in Ocular Pseudoexfoliation. Cureus. 2024 Jun 22;16(6):e62933. doi: 10.7759/cureus.62933. eCollection 2024 Jun. PMID 39050290
- [Background] Tomczyk-Socha M, Tomczak W, Winkler-Lach W, Turno-Krecicka A. Pseudoexfoliation Syndrome-Clinical Characteristics of Most Common Cause of Secondary Glaucoma. J Clin Med. 2023 May 21;12(10):3580. doi: 10.3390/jcm12103580. PMID 37240686
- [Background] Plateroti P, Plateroti AM, Abdolrahimzadeh S, Scuderi G. Pseudoexfoliation Syndrome and Pseudoexfoliation Glaucoma: A Review of the Literature with Updates on Surgical Management. J Ophthalmol. 2015;2015:370371. doi: 10.1155/2015/370371. Epub 2015 Oct 29. PMID 26605078